CLINICAL TRIAL: NCT01916369
Title: A Phase I Ascending Dose Safety Study Of Intramuscular CTX0E03 In Patients With Lower Limb Ischaemia
Brief Title: Safety Trial Of CTX Cells In Patients With Lower Limb Ischaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReNeuron Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN09-CP-0001; 2011-005810-13 (EudraCT Number)
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Fontaine Stage II, III or IV; Vascular disease; Cardiovascular diseases; Neural stem cell
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CTX DP (Experimental): Human neural stem cell product, single dose administered once only, increasing doses
  Interventions: Biological: CTX DP

INTERVENTIONS:
Biological: CTX DP — Single dose treatment consisting of 10 injections (20, 50 or 80 million cells) into the gastrocnemius muscle near to the damaged area
  Other Names: CTX0E03

SUMMARY:
The primary objective of the Phase I ascending dose trial is to investigate the safety and tolerability of intramuscular (gastrocnemius) injections of human neural stem cell product, CTX, in patients with peripheral arterial disease (Fontaine Stage II through IV). This trial is based on independent preclinical data from a leading academic research institution that has been submitted for publication. Inclusion of patients with Fontaine Stage II is justified as these patients have a lower incidence of background events and will facilitate distinction between events which are possibly intervention-related versus spontaneous events associated with underlying advanced atherosclerosis. The trial is designed to treat 9-18 patients and evaluate safety measures over a 12 month follow-up period.

DETAILED DESCRIPTION:
Design: The trial is a multi-centre open label, non-comparative, ascending dose safety study, using CTX cells to treat patients with lower limb ischaemia, with follow-up over 12 months.

Pre-treatment selection of patients: Men and women, aged >50 years with peripheral arterial occlusive disease (Fontaine Stage II through IV) of one leg or both, unsuitable for surgical re-vascularisation, an ankle/brachial pressure index (ABPI) of <0.9 or a toe/brachial index of <0.7. Women must be surgically sterile or more than 2 years past their last menstrual period and test negative for pregnancy.

Treatment: One patient will be treated at one time with a single dose of CTX cells. Three ascending doses (20, 50 or 80 million cells), allocated sequentially, will be tested in 9-18 patients (3 dose cohorts of 3-6 patients. All trial patients will receive 10 intramuscular injections of CTX DP into the gastrocnemius muscle of their ischaemic leg on a single occasion. In the event that both legs have peripheral arterial disease, the injections will be administered to the leg determined by the Investigator to have the more advanced/severe disease provided that leg has not already had surgical amputation of toes or above.

A minimum interval of 28 days will be observed between dosing the first and second patient and 7 days between dosing subsequent patients in a given cohort in order to assess the safety and tolerability of CTX DP at that dose. A further 3 patients may be added to any cohort (to a maximum of 18 of total treated patients) at the discretion of the Data Safety Monitoring Board (DSMB) if required to further clarify the safety profile). A minimum interval of 28 days will be observed between dosing the first and second patient and 7 days between dosing subsequent patients in a given cohort in order to assess the safety and tolerability of CTX DP at that dose.

Post-treatment follow-up: There will be 8 scheduled visits to the clinic for monitoring over the 12 month follow-up period.

End-points: The primary endpoint of the trial is safety, measured by numbers of relevant adverse events, health screening, physical examination (overall and of the treated limb), immunological response, amputation and concomitant medications in the first year after treatment.

Post-trial follow-up: Life-long annual follow-up to record any new cancer via national cancer registry or similar system or by Investigator or family practitioner (as permitted by competent authorities, ethics committees and informed consent).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent obtained from the patient.
* Peripheral arterial occlusive disease due to atherosclerosis (Fontaine stages II, III or IV) of one leg or both defined as
* Fontaine stage II: Intermittent claudication
* Fontaine stage III: Rest pain
* Fontaine stage IV: Ischaemic ulcer or (dry) gangrene
* Patients unsuitable for surgical re-vascularisation
* An ABPI of <0.9 or a toe/brachial index of <0.7
* Age >50 years
* Males or Females. Women must be surgically sterile or more than 2 years post their last menstrual period and with a negative pregnancy test.
* Smoker or non-smoker
* Diabetics and non-diabetics provided HbA1c <8% (or 64 mmol/mol)

Exclusion Criteria:

* Estimated survival of less than 6 months.
* Infection of the involved extremity manifested by fever, purulence, or severe cellulitis or active wet gangrenous tissue wound with exposed tendon or bone.
* Failed ipsilateral revascularisation procedure within 8 weeks prior to enrolment (defined as failure to restore adequate circulation, i.e., the procedure did not achieve an increase in ABPI of 0.15 or more, substantial improvement in Pulse Volume Recording, or clinical improvement).
* Previous amputation of the talus or above in the target limb.
* Planned major amputation within one month of planned date for injection of study medication (CTX DP).
* Anticoagulants including heparin, warfarin or analogues within the past month unless these can be discontinued per protocol for seven days prior to injection and two days post injection in the case of warfarin or one day prior to injection and two days post injection in the case of heparin or other anticoagulants.
* A history of deep vein thrombosis in either leg.
* Previous treatment with systemic growth pro-angiogenic factors or with stem-cell therapy.
* Ulcers from venous or neuropathic origin.
* Uncontrolled blood pressure defined as sustained systolic blood pressure ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg on repeated measures on different days.
* Acute cardiovascular events (e.g., myocardial infarction, stroke, recent coronary intervention) up to 6 months prior to enrolment.
* Previous or present history of malignant disease (except basal-cell carcinoma and cervical carcinoma in situ, which was removed without recurrence more than 5 years prior to enrolment).
* Body mass index >35.
* Previously diagnosed as clinically immune-compromised or taking systemic immunosuppressant medication.
* Patients taking sodium valproate for any indication within the past week.
* Organ transplant recipient.
* Inability to comprehend consent information or unlikely to comply with study requirements
* Participation in another study involving an Investigational Medicinal Product within the 3 months or 5 half-lives of the product (whichever is longer) prior to enrolment.
* Drug or alcohol abuse.
* Any other significant disease or abnormalities likely to impact study compliance or interpretation of the results. (If in doubt consult with the ReNeuron study monitor).
* Patients taking tamoxifen or analogues.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events | 12 months
  Monitoring of medical history, general physical examination, physical examination of the ipsilateral leg (inflammation, infection, swelling, tenderness, ulceration, gangrene), temperature, pulse rate and rhythm, ECG, blood pressure, full blood count, liver function tests, serum urea and electrolytes, creatine phosphokinase(muscle isoform), immunological response to CTX, amputation and concomitant medication.

CONTACTS AND LOCATIONS:
Overall Officials: Jill JF Belch, MBChB, Principal Investigator — Ninewells Hospital Dundee
Locations (1):
- Ninewells Hospital, Dundee, Scotland, United Kingdom

REFERENCES:
- [Derived] Stevanato L, Thanabalasundaram L, Vysokov N, Sinden JD. Investigation of Content, Stoichiometry and Transfer of miRNA from Human Neural Stem Cell Line Derived Exosomes. PLoS One. 2016 Jan 11;11(1):e0146353. doi: 10.1371/journal.pone.0146353. eCollection 2016. PMID 26752061